CLINICAL TRIAL: NCT01592734
Title: Efficacy and Tolerability of PEG-only Laxative for Fecal Impaction and Chronic Constipation in Children. A Controlled Double Blind Randomized Study vs a Standard PEG-EL Laxative
Brief Title: Efficacy and Tolerability of PEG-only Laxative for Fecal Impaction and Chronic Constipation in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Policlinico Umberto I (Other)
Collaborators: Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna (Other)
Responsible Party: Principal Investigator, Giovanni Di Nardo, MD, Azienda Policlinico Umberto I
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEG-P1
Record Dates: First submitted 2012-05-04; First posted 2012-05-07 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Constipation; Faecal Impaction
Keywords: chronic constipation; faecal impaction; PEG-only laxative
MeSH Terms: conditions — Constipation; Fecal Impaction | interventions — Polyethylene Glycols; Electrolytes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG-only (Experimental): Polyethylene glycol 4000 only (PEG-only).
  Interventions: Device: Polyethylene glycol
- PEG-EL (Active Comparator): Polyethylene glycol 3350 with electrolytes (PEG-EL).
  Interventions: Drug: Polyethylene glycol with electrolytes

INTERVENTIONS:
Drug: Polyethylene glycol with electrolytes — Constipation treatment: 1-4 sachets/day according to the patient age. 1 sachet contains 6.9 g PEG-EL. Treatment period: 4 weeks.
  Faecal impaction resolution: 4 sachets as initial dose and increasing 2 sachets a day until resolution or up to 7 days.
  Other Names: Movicol bambini
  Arms: PEG-EL
Device: Polyethylene glycol — Constipation: 0.7 g/kg/day in 2 divided doses for children of less than 20 kg. For children > 20 kg the daily dose was up to PEG 30 g daily. Treatment period: 4 weeks.
  Faecal impaction resolution: 1.5 g/kg/day in 2 doses until resolution or up to 6 days.
  Other Names: Onligol
  Arms: PEG-only

SUMMARY:
The aim of this study is to compare the efficacy, tolerability, acceptance and compliance of a PEG-only formulation compared to a reference PEG-EL formulation in resolving faecal impaction and in the treatment of chronic constipation

DETAILED DESCRIPTION:
Constipation is a very common complaint in childhood. Inadequate daily fiber intake, insufficient fluid intake, and withholding behavior are considered as factors leading to constipation.

Painful defecation is considered a common trigger to faecal retention wich leads to reabsorption of fluids and increase in the size and consistency of stools.

It is often necessary to use laxative therapy to achieve comfortable defecation. PEG-based laxatives are considered today the gold standard for treatment of constipation in children. PEG formulations differ for composition in inactive ingredients which may have an impact on acceptance, compliance and adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* out-patients children with diagnosis of functional constipation or have faecal impaction on medical history and physical examination

Exclusion Criteria:

* children with organic causes for defecation disorders, such as Hirschsprung disease, spina bifid, hypothyroidism, or other metabolic or renal abnormalities;
* Children receiving medication influencing gastrointestinal motility;
* Children with suspected gastrointestinal obstruction or stenosis

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Efficacy | 4 weeks of observation
  Stool frequency over the 4 weeks of treatment: daily recording of the number of stool on a patient diary card
Efficacy | 7 days
  Feacal impaction resolution

SECONDARY OUTCOMES:
Clinical tolerability | 4 weeks of observation
  Recording of all Adverse Events (AEs) occurred during the study
Acceptability | 4 weeks of observation
  Palatability and easy of taking the solution evaluated by a 5-points scale
Compliance | 4 weeks
  Percentage of patients who took more than 80% of the prescribed dose
Efficacy | 4 weeks
  Painfull stools, frequency of abdominal pain, frequency of soling episodes, use of stimulant laxatives by collection data on a patient diary card

REFERENCES:
- [Derived] Savino F, Viola S, Erasmo M, Di Nardo G, Oliva S, Cucchiara S. Efficacy and tolerability of peg-only laxative on faecal impaction and chronic constipation in children. A controlled double blind randomized study vs a standard peg-electrolyte laxative. BMC Pediatr. 2012 Nov 15;12:178. doi: 10.1186/1471-2431-12-178. PMID 23152962